CLINICAL TRIAL: NCT00354393
Title: Aggressive Multi-Modality Management of Malignant Pleural Mesothelioma
Brief Title: Combination Chemotherapy With or Without Surgery & Chemoradiotherapy in Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE-CCF-IRB-5179; P30CA043703 (NIH); CASE-CCF-IRB-5179 (Other: Internal IRB)
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma; sarcomatous mesothelioma; advanced malignant mesothelioma; epithelial mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Cisplatin; Methotrexate; Vinorelbine; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Induction Combination Chemotherapy (Experimental): Induction chemotherapy: Patients get MVP chemo. Treatment repeats every 28 days for 2 courses.
  Patients w/ unresectable disease may get up to 2 add'l courses of induction chemo. Patients requiring palliative radiotherapy or have PD are removed from study. Patients w/ resectable disease or sarcomatoid histology & T1-3, N1-2 disease w/ a CR or PR to induction chemo go to surgery.
  Surgery: Patients w/ extensive disease get palliative debulking pleurectomy and decortication & are taken off study. Other patients undergo a thoracotomy w/ extrapleural pneumonectomy & proceed to chemoradiotherapy.
  Chemoradiotherapy: At 6-10 weeks post-op, patients get 3-dimensional conformal or intensity-modulated radiotherapy once daily, 5 days a week, for 6 weeks. Patients receive cisplatin IV over 30-60 minutes days 1 & 22. Patients w/ responding disease proceed to adjuvant chemotherapy.
  Adjuvant chemotherapy: Patients get 2 more courses of MVP chemotherapy
  Interventions: Drug: Cisplatin; Drug: Methotrexate; Drug: Vinorelbine ditartrate; Procedure: Adjuvant therapy; Procedure: Conventional surgery; Procedure: Neoadjuvant Therapy; Radiation: 3-dimensional conformal radiation therapy; Radiation: Intensity-modulated radiation therapy

INTERVENTIONS:
Drug: Cisplatin
Drug: Methotrexate
Drug: Vinorelbine ditartrate
Procedure: Adjuvant therapy
Procedure: Conventional surgery
Procedure: Neoadjuvant Therapy
Radiation: 3-dimensional conformal radiation therapy
Radiation: Intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as methotrexate, vinorelbine, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Radiation therapy uses high-energy x-rays to kill tumor cells. Cisplatin may also make tumor cells more sensitive to radiation therapy. Giving chemotherapy and radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy with or without surgery and chemoradiotherapy works in treating patients with malignant pleural mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the response to induction combination chemotherapy comprising methotrexate, vinorelbine ditartrate, and cisplatin in patients with previously untreated malignant pleural mesothelioma.

Secondary

* Assess the tolerability and toxicity of this regimen in these patients.
* Determine relapse-free and overall survival of patients treated with induction combination chemotherapy with or without surgery and hemithoracic radiation.
* Assess the impact of induction combination chemotherapy on operability and surgical success.
* Evaluate the impact of these treatment regimens on quality of life.

OUTLINE:

* Induction chemotherapy: Patients receive MVP chemotherapy comprising cisplatin IV over 30-60 minutes on day 1 and vinorelbine ditartrate IV over 5-10 minutes and methotrexate IV over 5-30 minutes on days 8, 15, and 22. Treatment repeats every 28 days for 2 courses. Patients with unresectable disease may receive up to 2 additional courses of induction chemotherapy. Patients requiring palliative radiotherapy or who have progressive disease are removed from the study. Patients with resectable disease or sarcomatoid histology and T1-3, N1-2 disease with a complete or partial response to induction chemotherapy proceed to surgery.
* Surgery: Patients with extensive disease undergo palliative debulking pleurectomy and decortication and then are taken off study. All other patients undergo a thoracotomy with an extrapleural pneumonectomy and then proceed to chemoradiotherapy.
* Chemoradiotherapy: Beginning 6-10 weeks after surgery, patients undergo 3-dimensional conformal or intensity-modulated radiotherapy once daily, 5 days a week, for 6 weeks. Patients also receive cisplatin IV over 30-60 minutes on days 1 and 22. Patients with responding disease proceed to adjuvant chemotherapy.
* Adjuvant chemotherapy: Patients receive 2 additional courses of MVP chemotherapy as above.

Quality of life is assessed at baseline, after each course of induction chemotherapy, before surgery, and then every 3 months thereafter.

After completion of study therapy, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant pleural mesothelioma

  * Amenable to aggressive surgical resection, if deemed resectable

    * Patients with potentially resectable disease must have undergone mediastinoscopy to establish surgical stage

      * Resectable disease is defined as any of the following:

        * Epithelioid, mixed histology, or histology not otherwise specified with clinical stage I-III (T1-3, N0-2, M0) disease
        * Sarcomatoid histology with clinical stage I-III (T1-3, N0) disease
  * Intraperitoneal extension, contralateral thoracic extension, or distant metastases are eligible, but considered unresectable

    * Disease considered unresectable by any medical reason or if surgery was declined

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 3,000/mm³
* Platelet count > 100,000/mm³
* Creatinine ≤ 1.7 mg/dL
* Alkaline phosphatase < 2 times normal
* AST < 2 times normal
* Albumin > 3 g/dL
* Bilirubin < 2.0 mg/dL
* Patients must be available for and compliant with adequate long-term follow-up
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patients with resectable disease must have adequate pulmonary function to undergo surgery and radiotherapy
* No other active malignancies

PRIOR CONCURRENT THERAPY:

* No prior surgical resection, radiation therapy, chemotherapy, or immunotherapy for this cancer

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2002-08 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Best Response | After 2-4 cycles of induction chemotherapy (28 day cycle)
  Best response to chemotherapy after induction

SECONDARY OUTCOMES:
Tolerability and toxicity | After 2-4 cycles of induction chemotherapy (28 day cycle)
  Toxicity related to induction chemotherapy
Relapse free and overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first
  Time to relapse and overall survival
Assess Patient Quality of Life | Prior to initiation of each cycle of therapy, and every 3 months after completion of therapy until death, withdrawal or loss to follow up (Average 10 years)
  Patient Quality of Life during induction chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: David J. Adelstein, MD, Study Chair — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Shared on Physician Data Query